CLINICAL TRIAL: NCT03088787
Title: Feasibility of Continuous Noninvasive Finger Arterial Blood Pressure Measurement for Detection and Staging of Aortic Stenosis
Acronym: COaRt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, D.P.Veelo, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W17_072
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Aortic Stenosis, Calcific
MeSH Terms: conditions — Aortic Valve, Calcification of

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients for TAVR: Patients for TAVR
  Interventions: Device: Nexfin measuremtents

INTERVENTIONS:
Device: Nexfin measuremtents — There will be only observational recordings, no interevntion

SUMMARY:
The primary purpose of this study is electronic data collection of arterial pressure waveform signals in patients with Aortic Stenosis. The collected digital pressure waveform data will be used to assess the feasibility of using the arterial pressure signal as a decision support tool for early detection of aortic stenosis conditions. Furthermore we evaluate hemodynamic parameters before and after valve repair and its correlation with outcome.

ELIGIBILITY:
Inclusion Criteria:

* o Patients with severe senile degenerative aortic valve stenosis

  * Clinical team agrees on eligibility including assessment that TAVR is appropriate for the subject
  * Patients undergoing TAVR via the femoral approach
  * Patients who normally require a guiding catheter for central aortic pressure monitoring during the TAVR procedure
  * Patient must be 18 years old or older
  * Patient, or legally authorized representative, has given consent to be in the study
  * Patient height and weight are available prior to study
  * Ability to perform a Nexfin measurement at the left hand side.

Exclusion Criteria:

* o Patients with contraindications for placement of aortic catheter

  * Patients with mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation >3+).
  * Aortic valve is a congenital unicuspid or congenital bicuspid valve, or is noncalcified
  * Patients being treated with an intra-aortic balloon pump
  * Patients less than 40 kg in weight
  * Female patients of childbearing potential with a known pregnancy
  * Patient is currently participating in an investigational drug or another device study that clinically interferes with the study endpoints

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with aortic stenosis undergoing transcatheter aortic valve replacement (TAVR) procedures
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
the distinctive morphological characteristics of the aortic pressure waveform | During procedure and 4 hours after
  the distinctive morphological characteristics of the aortic pressure waveform

SECONDARY OUTCOMES:
changes in hemodynamic variables after TAVR and its influence on cardiac recovery. | during procedure and up to 6 weeks after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Veelo, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kho E, Schenk J, Vlaar APJ, Vis MM, Wijnberge M, Stam LB, van Mourik M, Jorstad HT, Hermanns H, Westerhof BE, Veelo DP, van der Ster BJP. Detecting aortic valve stenosis based on the non-invasive blood pressure waveform-a proof of concept study. Geroscience. 2024 Dec;46(6):5955-5965. doi: 10.1007/s11357-024-01136-w. Epub 2024 Mar 20. PMID 38509415
- [Derived] Schenk J, Kho E, Rellum S, Kromhout J, Vlaar APJ, Baan J, van Mourik MS, Jorstad HT, van der Ster BJP, Westerhof BE, Bruns S, Immink RV, Vis MM, Veelo DP. Immediate reduction in left ventricular ejection time following TAVI is associated with improved quality of life. Front Cardiovasc Med. 2022 Sep 16;9:988840. doi: 10.3389/fcvm.2022.988840. eCollection 2022. PMID 36187009